CLINICAL TRIAL: NCT05603299
Title: Establishing Clinical Utility Evidence to Support Coverage and Reimbursement for Venn Biosciences' DawnTM: A CPV® Randomized Controlled Trial
Brief Title: Establishing Clinical Utility Evidence to Support Coverage and Reimbursement for Venn Biosciences' Dawn Test
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study recruited no participants due to a pre-recruitment decision by the sponsor to not proceed. Factors considered included logistics, resources, and new research data.
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Venn Biosciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00062590
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The Control group treats their simulated patients using standard practice and have no introduction to the new test.
- Intervention Group 1 - Test Results Given (Experimental): Receiving educational materials describing the clinical validation and use cases of a predefined Dawn™ test and is given specific Dawn™ test results in Round 2 of CPV administration, whether they order the test or not.
  Interventions: Other: Educational Materials on the Dawn test
- Intervention Group 2 - Test Results Optional (Experimental): Receiving educational materials describing the clinical validation and use cases of a predefined Dawn™ test and is given specific Dawn™ test results in Round 2 of CPV administration, only if they choose to order the test.
  Interventions: Other: Educational Materials on the Dawn test

INTERVENTIONS:
Other: Educational Materials on the Dawn test — Receive educational materials and sample test results replicating what physicians would receive in the real-world market as they learn about the probability of IO therapy response from the Dawn™ test.
  Arms: Intervention Group 1 - Test Results Given; Intervention Group 2 - Test Results Optional

SUMMARY:
QURE will use its CPV technology in a randomized controlled trial to measure how InterVenn Biosciences diagnostic test changes clinical practice and improves patient outcomes.

DETAILED DESCRIPTION:
VennBio has developed a pioneering technology, Dawn™, a semi-quantitative assay using ultra-high-pressure-liquid chromatography, quantitative mass spectrometry (MS) that predicts the likelihood of a benefit from pembrolizumab (Keytruda®) or nivolumab (Opdivo®) plus ipilimumab (Yervoy®)), three of the most widely used immune checkpoint inhibitors currently available in the market. The Company's technology is powered by glycoproteomics and artificial intelligence (AI). The AI allows measuring of the glycoproteins and biological makeup of a patient. This combination of technology is meant for physicians to make the best decisions for patient outcomes in immuno-oncology (IO) therapies.

VennBio hopes to make Dawn™'s glycoproteomic solution widely available and is looking to accelerate the adoption of the test in patients with advanced/metastatic NSCLC. To make the test available to more patients, VennBio is looking for established, innovative approaches to gather high-quality prospective clinical utility data quickly. These data will be essential to increase access to the test and to gain coverage and reimbursement.

Accordingly, the proposed study will collect high-quality randomized controlled data from a nationally representative sample of practicing medical oncologists. The primary purposes of this study will be to 1) determine how these physicians currently choose therapy for advanced (i.e., locally advanced, unresectable, or metastatic) NSCLC patients, 2) ascertain if introducing the Dawn™ test will improve clinical decision-making, and 3) observe how the educational materials affect physician uptake of the Dawn™ test and treatment of their patients, particularly in assigning immunotherapy (e.g., IO monotherapy vs combination treatment with chemotherapy). Data from this study will investigate the best use case (type of patient) optimally served by Dawn™ testing (and thus the greatest clinical utility) and what physician characteristics (e.g., age, practice setting, training) and practice characteristics (e.g., multi-specialty, private practice, etc.) are associated with these practice changes.

QURE Healthcare is a team of clinicians and researchers that conducts randomized-controlled trials using Clinical Performance and Value (CPV®) patient simulations to generate high-quality clinical utility evidence. CPVs are QURE's scientifically-validated measurement tool, first described in the Journal of American Medical Association (JAMA) in 2000 and now used in scores of scientific investigations. In this research and derivative peer-reviewed publications, QURE's CPV studies efficiently measure clinical practice patterns among active physicians to determine if there is the value of new technologies to payers.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified medical oncologists for at least two years
* Averaging at least 20 hours per week of clinical and patient care duties over the last six months
* Routinely evaluate patients with advanced/metastatic NSCLC in their practice
* Prescribe IO therapies for their advanced/metastatic NSCLC patients
* Practice in either an academic, non-academic, or network hospital setting
* Practicing in the U.S.
* English speaking
* Access to the internet
* Informed, signed, and voluntarily consented to be in the study

Exclusion Criteria:

* Not board-certified in oncology
* Not English speaking
* Not averaging at least 20 hours per week of clinical and patient care duties over the last six months
* Not practicing in the U.S.
* No access to the internet
* Did not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-21 (Estimated); Primary Completion 2023-12-18 (Estimated); Study Completion 2023-12-18 (Estimated)

PRIMARY OUTCOMES:
CPV-measured clinical score difference | [6 months]
  Pre- and post-difference in the overall and the diagnostic and treatment quality scores between control physicians using standard of care diagnostic tools and intervention physicians using the Dawn™ test. In each CPV, participants' care recommendations are evaluated against evidence-based care scoring criteria which can sum from 0 to a high potential score of up to 100 percent in each domain, where higher scores mean better outcomes. The investigators will measure the overall change in the evidence-based physician behavior including physical exam, workup, diagnosis, and treatment of lung cancer in the CPV patient simulations.
CPV-measured cost difference | [6 months]
  Change in cost of related care for patients with lung cancer when comparing the control to the intervention group. (This cost is modeled in part by measuring differential rates of medical interventions selected by each arm and multiplying by average Medicare reimbursement rates for these interventions. The cost is also modeled by examining average per annum costs for patients suffering from lung cancer and multiplying by the percent of patients whose workup and interventions for cancer risks are significantly reduced following the intervention.)

SECONDARY OUTCOMES:
CPV-measured baseline clinical variation levels | [6 months]
  Participants completing the simulated cases, or CPVs, receive scores based upon the quality of care they provide. This measure will assess the baseline levels of variation in the care of pain patients among all participants, including by use case types. The investigators will measure the baseline levels of variation in the assessment, recognition, and management of lung cancer among all participants.
CPV-measured assessment of use case types | [6 months]
  The difference in the overall, and the diagnostic and treatment quality scores between control and intervention participants. Diagnostic and treatment scores are calculated as the percent correct on CPVs, and the overall score is an average score of the subcategory scores (percent correct). This will be examined for each of the use cases to determine in which case(s) CPV scores most improved.

CONTACTS AND LOCATIONS:
Overall Officials: John W Peabody, MD, PhD, Principal Investigator — QURE Healthcare